CLINICAL TRIAL: NCT01783327
Title: Teens-Connect: Preventive Psycho-education for Transitioning Teens With Diabetes
Acronym: TeensConnect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1112009416
Record Dates: First submitted 2013-01-28; First posted 2013-02-04 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Self care; Coping skills; Adolescent; Internet; Intervention Studies; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Chronic Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teens-Connect (Experimental): The Teens-Connect Program is an internet-based program that combines Managing Diabetes and TEENCOPE.
  Interventions: Behavioral: Teens-Connect
- Planet D (Active Comparator): Planet D is an internet program developed by the American Diabetes Association for children and adolescents with diabetes.
  Interventions: Behavioral: Planet D

INTERVENTIONS:
Behavioral: Teens-Connect — Teens-Connect combines Managing Diabetes and TEENCOPE. Managing Diabetes consists of 5 sessions on age-appropriate, educational content related to diabetes problem-solving and self-efficacy to improve self-management. TEENCOPE consists of 5 sessions designed to increase youth's sense of competence and mastery by retraining inappropriate or non-constructive coping styles and forming more positive styles and patterns of behavior. The program is highly interactive and youth can talk with each other on an online moderated discussion board. Youth will be asked to use the website at least twice per week for 4 weeks.
  Arms: Teens-Connect
Behavioral: Planet D — Planet D provides age-appropriate diabetes education on a variety of topics and social networking discussion boards on diabetes, food and exercise, personal interests, and diabetes camp. Planet D addresses emotions and self-management through education and social networking. Youth who register can also create a profile, upload and share pictures, identify favorite news and blog feeds as well as provide comments or tags to other members. Planet D has been online since 2007 and contains numerous diabetes-related articles geared toward youth as well as a secure message board. Youth will be asked to interact with the website twice a week for 4 weeks.
  Arms: Planet D

SUMMARY:
The purpose of this study is to evaluate the use of a state-of the art internet psycho-educational program in clinical practice (Teens-Connect), compared to use of a standard and widely available internet diabetes program for youth (Planet D™) in a mixed-method randomized clinical trial design.

DETAILED DESCRIPTION:
The aims are:

1. To evaluate the efficacy and cost-effectiveness of provider-prescribed Teens-Connect (TEENCOPE™+Managing Diabetes) in pediatric diabetes practice compared to prescription of Planet D™.

   The hypotheses to be studied are:
   1. Youth who participate in Teens-Connect will have better metabolic control (A1c) and quality of life (QOL) than those who participate in Planet D.
   2. These effects will be mediated by improvements in stress/coping, self-efficacy, diabetes problem-solving, and self-management.
   3. Teens-Connect prescribed by providers in diabetes clinics will be a cost-effective approach to reduce A1c and improve quality-adjusted life years (QALYs) for youth with T1D.
2. To compare the reach, efficacy, adoption, implementation, and maintenance (RE-AIM) of the two provider-prescribed psycho-educational internet programs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes for at least 6 months
* Age 11 to 14 years
* English-speaking
* Assent
* Parent/guardian consent to participate in study

Exclusion Criteria:

*Previous exposure to TEENCOPE and/or Managing Diabetes

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline hemoglobin A1c over 12 months | Baseline, 6 weeks, 6 months, 12 months
Change from baseline quality of life over 12 months | Baseline, 6 weeks, 6 months, 12 months

SECONDARY OUTCOMES:
Change from baseline coping/Stress over 12 months | Baseline, 6 weeks, 6 months, 12 months
  Coping/stress will be measured using the Perceived Stress Scale
Change from baseline self-efficacy over 12 months | Baseline, 6 weeks, 6 months, 12 months
  Self-efficacy will be assessed using the Self-efficacy for Diabetes Scale
Change from baseline problem-solving over 12 months | Baseline, 6 weeks, 6 months, 12 months
  Problem-solving will be assessed using the Self-Management of Diabetes-Adolescent (SMOD-A) questionnaire
Change from baseline self-management over 12 months | Baseline, 6 weeks, 6 months, 12 months
  Self-management will be assessed using the Self-care Inventory (SCI)
Costs | 6 months
  Costs will be assessed using financial and staff records
Change from baseline quality adjusted life years over 12 months | Baseline, 6 weeks, 6 months, 12 months
  Quality adjusted life years will be assessed using the Health Utilities Index Step 3 (Adolescent and Parent)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Grey, DrPH, Principal Investigator — Yale School of Nursing; Robin Whittemore, PhD, Principal Investigator — Yale School of Nursing
Locations (2):
- United States (2):
  - Yale University School of Nursing, New Haven, Connecticut
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania